CLINICAL TRIAL: NCT03361943
Title: Analysis of National Health and Nutrition Examination Survey (NHANES) 2003-2014 Data to Evaluate Trends in Sugar-sweetened Beverage (SSB) Intakes in Children
Brief Title: NHANES 2003-2014 and Sugar-sweetened Beverages in Children
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Michelle Mendez, Visiting Associate Professor, University of Pittsburgh
Other Study IDs: mendezssb1
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Sugar Sweetened Beverage Intakes in US Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study uses data from the NHANES surveys to evaluate trends in SSB intakes among US children. The goal was to determine whether recent declines in intake may have been less marked in the more vulnerable groups with a persistently high burden of obesity, including race/ethnic minorities and low-income groups.

DETAILED DESCRIPTION:
Recent studies suggest sugar-sweetened beverage (SSB) consumption has been declining among US children 2-18y. However, most studies focus on changes in mean intake and little is known about trends in the high SSB consumers who are most at risk of excess weight gain. There is also limited understanding of whether and how these changes over time may have influenced disparities in intake among vulnerable groups of children with persistently high levels of obesity, including children from low-income households, and several race-/ethnic minorities.

This analysis of six cycles of US National Health and Nutrition Examination Survey (NHANES) dietary surveillance data from 2003-2014 examined shifts over time in SSB intake at both the median and 90th percentile among US children. The study evaluated the extent to which disparities in intake of total SSBs, as well as major SSB subtypes (regular sodas, fruit drinks and other), may have persisted in vulnerable groups, for both median and "heavy" intake. The analysis presents data for three age groups: 2-5y, 6-11y and 12-18y by gender, and focus on three race-ethnic groups: Non-Hispanic White, Non-Hispanic Black, and Mexican-American. Household income is used as the primary socioeconomic status variable.

ELIGIBILITY:
Inclusion Criteria:

* All U.S. children aged 2-18y in US NHANES diet surveys from 2003-2014

Exclusion Criteria:

* missing socio-economic data: parental education or household income as a percentage of the Federal Poverty Level; n=1841
* missing or implausible dietary data, defined as: energy intake of zero kcal or more than four standard deviations beyond individual estimated energy requirements, or no report on whether data represents usual intake (more, same or less than usual); n=236

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 17,579 children aged 2-18 years in US NHANES dietary surveys from 2003-2014 with household socioeconomic data
Sampling Method: Probability Sample
Enrollment: 17579 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Sugar Sweetened Beverage Intake in Children | 2003-2014
  All non-alcoholic, non-diet beverages sweetened with sugars of any type, either as purchased or added after purchase